CLINICAL TRIAL: NCT03126825
Title: Clinical Evaluation of the SpatialNR Noise Reduction Algorithm
Brief Title: CLEAR Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5606
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional CI (Other): The conventional CI group will receive the noise reduction on and off signal processing test programs. This is a within subject repeated measures design, so all subjects will receive the same testing but in a counterbalanced order.
  Interventions: Device: CP910/CP920 with noise reduction on; Device: CP910/CP920
- Hybrid CI (Other): The Hybrid CI group will receive the noise reduction on and off signal processing test programs. This is a within subject repeated measures design, so all subjects will receive the same testing but in a counterbalanced order.
  Interventions: Device: CP910/CP920 with noise reduction on; Device: CP910/CP920

INTERVENTIONS:
Device: CP910/CP920 with noise reduction on — This intervention uses the approved Nucleus 6 system (CP910/CP920 and accessories) but adds the investigational noise reduction algorithm.
Device: CP910/CP920 — The approved CP910 or CP920 Sound Processor.

SUMMARY:
Acute in-booth assessment of a new noise reduction algorithm with cochlear implant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Conventional CI subject aged twelve years of age or older, or Hybrid subject aged 18 years or older
2. Recipient of a CI500 Series (CI512 or CI522) or CI24RE Series (CI24REH or CI422) cochlear implant
3. At least three months CI experience in ear to be assessed
4. At least three months experience with the CP810,CP920 or CP910 sound processor
5. Fluent speaker in the local language used to assess clinical performance
6. Open-set speech perception ability
7. Use of or eligibility for hybrid acoustic component (hybrid population only)

Exclusion Criteria:

1. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations that are inherent to the investigational device
2. Unwillingness or inability of the candidate to comply with all investigational requirements
3. Additional handicaps that would prevent or restrict participation in the audiological evaluations or that would affect the scientific integrity of the study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-08-13 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
CNC words | 3 months
  CNC words in quiet will be used to assess whether the investigational noise reduction algorithm performs no worse than the approved Nucleus 6 defaults.
SRT sentences | 3 months
  SRT sentences in noise will be used to assess whether the investigational noise reduction algorithm performs no worse than the approved Nucleus 6 defaults.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Brinson, Phd, Study Director — Head of Global Clinical Affairs
Locations (2):
- Australia (2):
  - Cochlear Limited Sydney, Sydney, New South Wales
  - Cochlear Limited Melbourne, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
Currently no plan to make IPD available to other researchers.